CLINICAL TRIAL: NCT00165750
Title: Correlation Between Regional Brain Volume and Response to Donepezil Treatment in AD Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of patients to enroll.
Sponsor: Eisai Korea Inc. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AS-019 (EKI-5-003)
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: DONEPEZIL HYDROCHLORIDE

INTERVENTIONS:
Drug: DONEPEZIL HYDROCHLORIDE — One 5mg table, once daily. (After 4 weeks treatment, the dose can be increased 10mg once daily.)
  Other Names: Aricept

SUMMARY:
This study investigate the relationship between regional brain volume measured by MRI and donepezil treatment response in patients with Alzheimer's Disease.

ELIGIBILITY:
Inclusion criteria:

1. Over 60 years old.
2. Probable or possible Alzheimer's Disease according to the DSM-IV and NINCDS-ADRDA.
3. MMSE score of 10~24, CDR of 1~2.
4. Patients didn't take acetylcholinesterase inhibitors 4 weeks before screening.
5. Permitted drugs: antipsychiatric drug for BPSD, antidepression drug, tranquilizer, treatment drug for physical disease for example hypertension.

Exclusion criteria:

1. Uncontrolled by donepezil because of adverse events.
2. No longer continuing treatment of donepezil for refuse, drug-drug interaction etc.
3. If they have taken concomitant medication which were not allowed.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-03; Primary Completion 2008-08 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
MRI, ADAS-cog | 0, 12, 24 weeks

SECONDARY OUTCOMES:
ADL, BPSD, CDR-SB, ZBI, GHQ, CIBIC plus | 0, 12, 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jihee Mun, Study Director — Eisai Korea Inc.
Locations (1):
- Cheonnam University Hospital, Gwangju, Gwangju, South Korea